CLINICAL TRIAL: NCT01573221
Title: Stroke and PMSI Evaluation of the Sensitivity and Specificity
Brief Title: Stroke and PMSI (Medicalisation Information Systems Programm)
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: GiroudPHRCN2010
Record Dates: First submitted 2012-04-04; First posted 2012-04-09 (Estimated); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- stroke

SUMMARY:
Evaluation of the sensitivity and specificity of PMSI to identify the burden of stroke in France,from 2500 cases

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of stroke in the hospital activity board

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospitalized stroke
Sampling Method: Probability Sample
Dates: Start 2011-07 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurice GIROUD, Principal Investigator — Centre Hospitalier Universitaire Dijon
Locations (2):
- France (2):
  - CHU Dijon, Dijon
  - CHU Grenoble, Grenoble